CLINICAL TRIAL: NCT02262312
Title: Iron Overload and Transient Elastography in Patients With Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-402
Record Dates: First submitted 2014-09-18; First posted 2014-10-13 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients with myelodysplastic syndrome: Patients with myelodysplastic syndrome among these include also patients with chronic myelomonocytic leukemia with myelodysplasia, patients with acute myeloid leukemia progressed from myelodysplastic syndrome and patients with myelodysplastic/myeloproliferative neoplasm, unclassifiable
  Interventions: Other: Transient elastography

INTERVENTIONS:
Other: Transient elastography — All patients will have a transient elastography performed as a measure of liver stiffness.
  Other Names: Fibroscan; Liver stiffness measurements

SUMMARY:
Patients with myelodysplastic syndrome (MDS) have an ineffective hemopoiesis and often suffer from anemia. This can lead to red blood cell transfusion dependency and iron overload. Iron overload can affect the liver and lead to liver fibrosis and worst case cirrhosis. Ferritin is usually used to monitor the iron overload. In this study MDS patients will have a transient elastography performed which measures the liver's stiffness. The purpose is to investigate whether liver stiffness measurements are coherent to ferritin levels.

DETAILED DESCRIPTION:
Transient elastography is noninvasive and has no side effects. No liver biopsy will be performed due to serious side-effects and risks in this patientgroup.

The results of the transient elastography will be compared to the patient's ferritin levels and the numbers of months the patients have had MDS to find out if there is a correlation. Furthermore we will compare the liver stiffness measurements in the patients with higher ferritin levels to those who have lower ferritin levels. We will also compare the liver stiffness measurements in patients who are red blood cell transfusion dependent compared to those who are red blood cell transfusion independent. We will also compare liver stiffness measurements in the patients with a high alanine aminotransferase (ALAT) compared to those with normal ALAT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a bone marrow describing myelodysplasia

Among these:

* Patients with myelodysplastic syndrome (MDS)
* Patients with acute myeloid leukemia (AML) transformed from MDS
* Patients with chronic myelomonocytic leukemia (CMML) with dysplasia
* Patients with myelodysplastic/myeloproliferative neoplasm, unclassifiable

Exclusion Criteria:

Body mass index (BMI) of 30 or higher than 30

- History with other known liver diseases

Among these:

* Patients with chronic viral hepatitis C infection
* Patients with chronic viral hepatitis B infection
* Patients with alcoholic liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myelodysplastic syndrome among these include also patients with chronic myelomonocytic leukemia with myelodysplasia, patients with acute myeloid leukemia progressed from myelodysplastic syndrome and patients with myelodysplastic/myeloproliferative neoplasm, unclassifiable.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Liver stiffness | Transient elastography (Fibroscan) 5 minutes
  Liver stiffness is measured in kilopascal (kPa)
Iron overload: Ferritin | Blood samples 5 minutes
  Ferritin is measured in micrograms per liter

SECONDARY OUTCOMES:
Disease period | Information regarding time of diagnosis will be obtained retrospectively
  Period of disease will be calculated in months
Red blood cell transfusion dependency | Information regarding transfusion will be obtained retrospectively
  Transfusion dependency will be defined as having at least one red blood cell transfusion every other eight weeks over a period of four months prior to the date of the fibroscan. Red blood cell dependency will be either "yes" or "no"
Liver inflammation: Alanine aminotransferase | Blood samples 5 minutes
  Alanine aminotransferase is measured in units per liter

CONTACTS AND LOCATIONS:
Overall Officials: Klas Raaschou-Jensen, Principal Investigator — Consultant at department of hematology
Locations (1):
- Department of hematology Roskilde hospital, Roskilde, Roskilde, Denmark